CLINICAL TRIAL: NCT05646979
Title: The Effect of Emotional Freedom Techniques on Anxiety, Surgical Fear and Traumatic Birth Perception of Pregnant Women Who Will Have a Planned Caesarean Section: A Randomised Controlled Study
Brief Title: The Effect of Emotional Freedom Technique Applied Before Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sinem GUVEN Santur, Pirincipal İnvestigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Inonu Universty, Malatya
Record Dates: First submitted 2022-12-04; First posted 2022-12-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section; Emotional Regulation; Surgery; Traumatic Birth
Keywords: Cesarean section; Emotional freedom technique; Surgery fear; Traumatic birth perception
MeSH Terms: conditions — Emotional Regulation; Birth Injuries

STUDY DESIGN:
Intervention Model Description: The randomized experiment was designed as a control study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): EFT application will be applied to the women in the experimental group who will have a cesarean section at 32-38 weeks of gestation.
  Interventions: Behavioral: EFT group
- Control group (No Intervention): Women in the control group who will have a cesarean section at 32-38 weeks of gestation will not be interfered with.

INTERVENTIONS:
Behavioral: EFT group — EFT protocol will be applied to the women in the experimental group who will have a cesarean section at 32-38 weeks of gestation.
  Arms: Experimental group

SUMMARY:
Since all the follow-up and care of the pregnant during the prenatal period are carried out by the midwives, the care provided by the midwives to the women during the prenatal period plays a key role for the woman to have a comfortable and healthy pregnancy. Midwives should take psychological approaches in order to reduce the negative feelings of women before cesarean section. Considering all these, it is thought that Emotional Freedom Technique, which does not require any invasive intervention, is inexpensive and easy to apply, will contribute to women's feeling better by reducing pre-cesarean anxiety, surgical fear and traumatic birth perception.

DETAILED DESCRIPTION:
Although childbirth is a normal physiological event for the female body, it causes stress for the woman and brings with it many risks. Cesarean section, which is one of the birth types; It is a surgical procedure that enables delivery to occur through an incision made on the abdominal wall and uterus of the mother. Although the cesarean rate recommended by the World Health Organization (WHO) is 15%, the rate of cesarean section in our country is 52.1% according to the Turkey Demographic and Health Survey.

Every surgical procedure to be performed, the decision of surgery and the waiting period may cause anxiety in individuals. Anxiety and fear experienced before surgery; It can cause individuals to experience uneasiness, restlessness and dissatisfaction due to the uncertainty they are in. Preoperative pain, fear of death, the thought that the body will be harmed and suffering, fear of losing consciousness and control due to anesthesia, and the uncertainty associated with anesthesia may cause fear of surgery. Anxiety before cesarean section is multifaceted, and it has been reported that the pregnancy process increases anxiety. In studies, it was determined that the anxiety level of mothers before cesarean section was high. The extreme degree of anxiety and fear plays a very important role in the formation of traumatic perception towards birth.

Many methods are used to reduce negative emotions in the prenatal period. Emotional Freedom Technique (EFT), which is one of these methods, is a method used to resolve emotional blockages in the energy body of the person. EFT aims to reveal all the points where there is a possibility of negative emotion experienced in the past and stuck in a part of the body. By focusing on the emotions that negatively affect the person in EFT, the energy flow is regulated with stimulations often made by touch. When administered to pregnant women, it may contribute to a decrease in post-traumatic stress disorder and to reduce the level of anxiety and fear.

Since all the follow-up and care of the pregnant during the prenatal period are carried out by the midwives, the care provided by the midwives to the women during the prenatal period plays a key role for the woman to have a comfortable and healthy pregnancy. Midwives should take psychological approaches in order to reduce the negative feelings of women before cesarean section. Considering all these, it is thought that EFT, which does not require any invasive intervention, is inexpensive and easy to apply, will contribute to women's feeling better by reducing pre-cesarean anxiety, surgical fear and traumatic birth perception.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* at 32-38 weeks of gestation,
* Cesarean delivery planned,
* Not carrying any risk factors (preeclampsia, IUGG, premature rupture of membranes, getational diabetes, etc.) during pregnancy,
* Single pregnancy,
* Not having any problems (such as fetal anomaly, intrauterine growth retardation) related to the health of the fetus,
* Pregnant women who do not have conditions such as infection, wound, scar in the tapping areas.

Exclusion Criteria:

* Diagnosing a risky pregnancy during the research process,
* Participant's unwillingness to continue with the EFT protocol

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Experience- (SUE) | Each participant will be evaluated for 1 week.
  The negative 10 feel the greatest pain, disappointment, fear, stress, sadness, or discomfort imaginable. When it reaches Positive 10, the client feels very different and wonderful. The meanings of the ratings in this range change gradually. The scale has no cutoff score. It is interpreted according to the mean of the scores and its relevance to other variables.

SECONDARY OUTCOMES:
Traumatic Birth Perception Scale | It will be applied as a post-test 1 week after it is applied as a pre-test to the pregnants between 32-38 weeks included in the study.
  The scale consists of a total of 13 questions covering thoughts and feelings such as anxiety, fear and anxiety that the woman feels when she thinks about the concept of birth. For each problem, a score is given from 0 to 10, whether I'm afraid or afraid. The lowest and highest scores that can be obtained from the scale are 0 and 130. According to the total mean score of the scale, the 0-26 score range is "very low", the 27-52 score range is "low", the 53-78 score range is "moderate", the 79-104 score range is "high", and the 105-130 score range is "very high" indicates the perception of traumatic birth.
Surgical Fear Scale | It will be applied as a post-test 1 week after it is applied as a pre-test to the pregnants between 32-38 weeks included in the study.
  The scale is in 11-point Likert type, consists of 8 questions and scores between 0 and 10. The scale, each of which consists of 4 items, consists of two sub-dimensions measuring short-term fears and long-term fears related to the source of fear. Items 1 to 4 in the scale measure the fear of short-term results of surgery, while items 5 to 8 measure the fear of long-term results. The items in the scale are evaluated as "0: I am not afraid at all" and "10: I am very afraid".
State anxiety scale | It will be applied as a post-test 1 week after it is applied as a pre-test to the pregnants between 32-38 weeks included in the study.
  The State Anxiety Scale is an individual's at a certain moment and under certain conditions; It requires him to describe how he feels. The emotions and behaviors expressed in the inventory items are indicated by choosing one of the options "(1) Not at all, (2) A little, (3) A lot and (4) Completely" according to the severity of such experiences. The total score obtained can vary between 20 and 80.
Demographic Descriptive Data | It will be obtained in 1 month at the beginning of the research.
  Pregnant information form prepared by the researcher in line with the literature, socio-demographic (pregnant woman's age, education and employment status, income status, family type and place of residence), obstetric (current gestational week and pregnancy history), psycho-social and medical history (desire for pregnancy) status, whether there is a chronic disease) consists of questions.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Karataş Okyay, Principal Investigator — https://akademik.ksu.edu.tr/Default.aspx?kod=CfTMEAi69foG7wFizm48ztSNEmgmVjdANJTT1Xcj9gA=; Zeliha Özşahin, Study Director — https://avesis.inonu.edu.tr/zeliha.ozsahin/bilimselfaaliyetler
Locations (1):
- Malatya Training and Research Hospital, Malatya, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In the research, data collection forms will be filled by face-to-face interview method. Data will be collected with Personal Information Form, State Anxiety Scale (STAI-I), Surgical Fear Scale, Traumatic Birth Perception Scale (TDAS) and Subjective Units of Experience (SUE) Scale.